CLINICAL TRIAL: NCT00628745
Title: Transthyretin Amyloidosis Outcomes Survey (THAOS): A Global, Multi-Center, Longitudinal, Observational Survey of Patients With Documented Transthyretin Gene Mutations or Wild-Type Transthyretin Amyloidosis.
Brief Title: Transthyretin Amyloidosis Outcome Survey (THAOS)
Acronym: THAOS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461001; FX-R-001 (Other: Alias Study Number); THAOS (Other: Alias Study Number)
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Transthyretin Gene Mutations; Transthyretin Amyloidosis
Keywords: TRANSTHYRETIN; AMYLOIDOSIS; TRANSTHYRETIN AMYLOIDOSIS; Transthyretin amyloid cardiomyopathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational
  Interventions: Other: None. Observational Study.

INTERVENTIONS:
Other: None. Observational Study.

SUMMARY:
THAOS is a global, multi-center, longitudinal observational survey open to all patients with transthyretin amyloidosis (ATTR), including ATTR-PN (polyneuropathy), ATTR-CM (cardiomyopathy) and wild-type ATTR-CM. It is open-ended with a minimum duration of 10 years. Patients will be followed as long as they are able to participate. The principal aims of this outcome survey are to better understand and characterize the natural history of the disease by studying a large and heterogenous patient population. Survey data may be used to develop new treatment guidelines and recommendations, and to inform and educate clinicians about the management of this disease.

DETAILED DESCRIPTION:
n/a NA

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria to be eligible for inclusion into THAOS:

1. Evidence of a personally signed and dated informed consent document indicating that the participant (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
2. Males and females greater than or equal to 18 years of age.
3. Confirmed genotyped TTR mutation with or without a diagnosis of hereditary or wild-type ATTR amyloidosis. Confirmation of ATTRwt amyloidosis will be determined by genotyped confirmation that patient does not possess a known mutation in TTR gene (ie, is a carrier of wild-type allele only) via genetic testing and one of the following set of criteria (a, b, or c):

   1. Presence of amyloid in cardiac biopsy tissue confirmed as TTR amyloid by mass spectrometry or immunohistochemistry; or
   2. Evidence of cardiac involvement by echocardiogram as defined by left ventricle wall thickness of >12 mm, and presence of amyloid in non-cardiac tissue confirmed as TTR amyloid by mass spectrometry or immunohistochemistry; or
   3. Evidence of cardiac involvement by echocardiogram as defined by left ventricle wall thickness of >12 mm, and presence of amyloid in cardiac tissue indirectly confirmed by scintigraphy with a "bone seeking tracer" eg, 99mTC-DPD [99mTC-3,3-diphosphono-1,2-propano-dicarboxylic acid], 99mTC- PYP [Pyrophosphate], and 99mTC-HMDP [hydroxymethylene diphosphonate] with Perugini grade greater than or equal to 2.

Exclusion Criteria

Patients meeting any of the following will not be included in the study:

1. Patient has evidence of primary (light chain) or secondary amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with confirmed hereditary or wild-type ATTR amyloidosis (inclusive of ATTR-PN and ATTR-CM) and those with TTR gene mutations without a diagnosis of ATTR amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 6718 (Actual)
Dates: Start 2008-01-04 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (112):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California - San Francisco, UCSF Department of Neurology, San Francisco, California
  - Office of Sponsored Research, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - UC Denver, Aurora, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - UHealth Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - UHealth Plantation, Plantation, Florida
  - Clinical Trials Unit, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center IRB, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Centre, Oak Lawn, Illinois
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cardiology Clinic at Montefiore Hutchinson Campus, The Bronx, New York
  - Montefiore Medical Center-Jack D. Weiler Hospital, The Bronx, New York
  - Congestive Heart Failure Clinic, The Bronx, New York
  - Montefiore Moses Division, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio University College of Medicine, Columbus, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Peters Township Health and Wellness Pavillion, McMurray, Pennsylvania
  - Penn Presbyterian Medical Center-University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Admin, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavillion, Wexford, Pennsylvania
  - IRB, Nashville, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - The University of Utah Health Sciences Center, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano de Buenos Aires (HIBA), Buenos Aires
  - FLENI, Buenos Aires
  - Instituto De Investigaciones Medicas Dr Alfredo Lanari, Buenos Aires
- Afdeling Klinische Cardiologie, O&N I, Leuven, Belgium
- Brazil (2):
  - Hospital Universitário Clementino Fraga Filho -HUCFF Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Instituto Dante Pazzanese De Cardiologia, São Paulo
- Alexandrovska University Hospital Clinic of Neurology, Sofia, Bulgaria
- Canada (3):
  - University of Alberta Foothills Medical Centre, Calgary, Alberta
  - Toronto General Hospital-University Health Network, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Cyprus Institute of Neurology and Genetics, Nicosia, Cyprus
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- France (7):
  - CHU de Bicetre, Cedex
  - Hopital Louis Pasteur, Colmar
  - CHU Henri Mondor, Créteil
  - Chu De Fort De France, Fort de France
  - CHRU de Lille, Hopital Claude Huriez, Lille
  - Hopital Salengro - CHRU de Lille, Lille
  - CHU de Toulouse - Hopital Rangueil, Toulouse
- Germany (7):
  - University Hospital of RWTH Aachen, Aachen
  - Charite CAmpus Rudolf-Virchow-Klinikum, Berlin
  - Medical University of Heidelberg, Heidelberg
  - Johann-Gutenberg-Universität, Mainz
  - University Medical Center, Johannes Gutenberg-University Mainz, Mainz
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz KöR, Mainz
  - Universitatsklinikum Muenster - Transplant Hepatology, Münster
- Israel (2):
  - Wolfson Medical Center, Holon
  - Sheba Medical Center, Ramat Gan
- Italy (8):
  - Comitato Etico Indipendente dell Azienda, Bologna
  - Azienda Ospedaliero-Universitaria di Careggi, Florence
  - AOU Policlinico G. Martino - Messina - Comitato Etico Scientifico, Messina
  - AOU Policlinico G. Martino - Messina - Dr. Vita, Messina
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Pavia - Prof. Merlini, Pavia
  - Comitato di Bioetica della Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio Per La Ricerca Medica E Di Sanita Pubblica (Ftgm), Pisa
  - Fondazione Policlinico Gemelli - Universita Cattolica del Sacro Cuore, Roma
- Japan (3):
  - Shinshu University School of Medicine, Matsumoto, JP
  - Chiba University Hospital, Chiba
  - Kumamoto University, Kumamoto
- University Malaya Medical Centre (UMMC), Kuala Lumpur, Kuala Lumpur, Malaysia
- Instituto Nacional de Ciencia Medicas y Nutricion Salvador Zubiran, Distrito Federal, Mexico
- University Medical Center Groningen, Groningen, Netherlands
- Portugal (4):
  - Centro Hospitalar Do Alto Ave, Epe, Guimarães
  - Centro Hospitalar Lisboa Norte (CHLN) EPE - Hospital de Santa Maria, Lisbon
  - Hospital Santa Maria, Lisbon
  - Unidade Clinica de Paramiloidose-Centro Hospitalar Porto,EPE-Hospital Geral Santo Antonio, Porto
- Institutul De Cardiologie Prof. Dr. C. C. Iliescu Spitalului Fundeni, Bucharest, Romania
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- South Korea (2):
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (9):
  - Hospital Universitario Donostia, Gipuzkoa - SanSebastian, Donostia
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Institut Clinic de Nefrologia i Urologia - ICNU, Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital de Rehabilitacion y Traumatologia Virgen de las Nieves, Granada
  - Hospital Juan Ramon Jimenez, Huelva
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Son Llàtzer, Palma de Mallorca
- Sweden (3):
  - Piteå Älvdals Hospital, Piteå
  - Karolinska University Hospital, Huddinge, Stockholm
  - Umeå University Hospital, Umeå
- National Taiwan University Hospital, Taipei, Taiwan
- Istanbul University,Istanbul Faculty of Medicine,Department of Neurology, Istanbul, Turkey (Türkiye)
- Cleveland Clinic Abu Dhabi LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wixner J, Dispenzieri A, Amass L, Carlsson M, Riley S, Powers E, Kelly JW. A real-world study of tafamidis in people with transthyretin amyloid cardiomyopathy (ATTR-CM) with heart and nerve symptoms: a plain language summary. Future Cardiol. 2025 Nov 25:1-13. doi: 10.1080/14796678.2025.2583805. Online ahead of print. PMID 41292260
- [Derived] Wixner J, Dispenzieri A, Amass L, Carlsson M, Riley S, Powers E, Kelly JW; THAOS investigators. Survival in a Contemporary, Real-World Cohort of Patients with Mixed-Phenotype Transthyretin Amyloid Cardiomyopathy Treated with Tafamidis: An Analysis from THAOS. Cardiol Ther. 2025 Dec;14(4):583-599. doi: 10.1007/s40119-025-00421-9. Epub 2025 Jul 9. PMID 40632476
- [Derived] Mora-Ayestaran N, Dispenzieri A, Kristen AV, Maurer MS, Diemberger I, Drachman BM, Grogan M, Gupta P, Glass O, Amass L, Garcia-Pavia P; THAOS Investigators. Age- and Sex-Related Differences in Patients With Wild-Type Transthyretin Amyloidosis: Insights From THAOS. JACC Adv. 2024 Jul 12;3(8):101086. doi: 10.1016/j.jacadv.2024.101086. eCollection 2024 Aug. PMID 39105117
- [Derived] Garcia-Pavia P, Kristen AV, Drachman B, Carlsson M, Amass L, Angeli FS, Maurer MS; THAOS investigators. Survival in a Real-World Cohort of Patients With Transthyretin Amyloid Cardiomyopathy Treated With Tafamidis: An Analysis From the Transthyretin Amyloidosis Outcomes Survey (THAOS). J Card Fail. 2025 Mar;31(3):525-533. doi: 10.1016/j.cardfail.2024.06.003. Epub 2024 Jun 21. PMID 38909877
- [Derived] Gentile L, Diemberger I, Plante-Bordeneuve V, Mazzeo A, Dori A, Luigetti M, Di Paolantonio A, Dispenzieri A, Grogan M, Waddington Cruz M, Adams D, Inamo J, Kristen AV, Lino Cirami C, Chapman D, Gupta P, Glass O, Amass L. Phenotypic characteristics of F64L, I68L, I107V, and S77Y ATTRv genotypes from the Transthyretin Amyloidosis Outcomes Survey (THAOS). PLoS One. 2024 Jan 19;19(1):e0292435. doi: 10.1371/journal.pone.0292435. eCollection 2024. PMID 38241252
- [Derived] Gonzalez-Moreno J, Dispenzieri A, Grogan M, Coelho T, Tournev I, Waddington-Cruz M, Wixner J, Diemberger I, Garcia-Pavia P, Chapman D, Gupta P, Glass O, Amass L; THAOS investigators. Clinical and Genotype Characteristics and Symptom Migration in Patients With Mixed Phenotype Transthyretin Amyloidosis from the Transthyretin Amyloidosis Outcomes Survey. Cardiol Ther. 2024 Mar;13(1):117-135. doi: 10.1007/s40119-023-00344-3. Epub 2023 Dec 20. PMID 38117424
- [Derived] Gentile L, Coelho T, Dispenzieri A, Conceicao I, Waddington-Cruz M, Kristen A, Wixner J, Diemberger I, Gonzalez-Moreno J, Cariou E, Maurer MS, Plante-Bordeneuve V, Garcia-Pavia P, Tournev I, Gonzalez-Costello J, Duarte AG, Grogan M, Mazzeo A, Chapman D, Gupta P, Glass O, Amass L; THAOS investigators. A 15-year consolidated overview of data in over 6000 patients from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Orphanet J Rare Dis. 2023 Nov 10;18(1):350. doi: 10.1186/s13023-023-02962-5. PMID 37946256
- [Derived] Coelho T, Conceicao I, Waddington-Cruz M, Keohane D, Sultan MB, Chapman D, Amass L; THAOS investigators. A natural history analysis of asymptomatic TTR gene carriers as they develop symptomatic transthyretin amyloidosis in the Transthyretin Amyloidosis Outcomes Survey (THAOS). Amyloid. 2022 Dec;29(4):228-236. doi: 10.1080/13506129.2022.2070470. Epub 2022 Jun 22. PMID 35730447
- [Derived] Dispenzieri A, Coelho T, Conceicao I, Waddington-Cruz M, Wixner J, Kristen AV, Rapezzi C, Plante-Bordeneuve V, Gonzalez-Moreno J, Maurer MS, Grogan M, Chapman D, Amass L; THAOS investigators. Clinical and genetic profile of patients enrolled in the Transthyretin Amyloidosis Outcomes Survey (THAOS): 14-year update. Orphanet J Rare Dis. 2022 Jun 18;17(1):236. doi: 10.1186/s13023-022-02359-w. PMID 35717381
- [Derived] Campbell CM, LoRusso S, Dispenzieri A, Kristen AV, Maurer MS, Rapezzi C, Lairez O, Drachman B, Garcia-Pavia P, Grogan M, Chapman D, Amass L; THAOS investigators. Sex Differences in Wild-Type Transthyretin Amyloidosis: An Analysis from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Cardiol Ther. 2022 Sep;11(3):393-405. doi: 10.1007/s40119-022-00265-7. Epub 2022 May 18. PMID 35583798
- [Derived] Barroso FA, Coelho T, Dispenzieri A, Conceicao I, Waddington-Cruz M, Wixner J, Maurer MS, Rapezzi C, Plante-Bordeneuve V, Kristen AV, Gonzalez-Duarte A, Chapman D, Stewart M, Amass L; THAOS investigators. Characteristics of patients with autonomic dysfunction in the Transthyretin Amyloidosis Outcomes Survey (THAOS). Amyloid. 2022 Sep;29(3):175-183. doi: 10.1080/13506129.2022.2043270. Epub 2022 Apr 22. PMID 35451899
- [Derived] Nativi-Nicolau J, Siu A, Dispenzieri A, Maurer MS, Rapezzi C, Kristen AV, Garcia-Pavia P, LoRusso S, Waddington-Cruz M, Lairez O, Witteles R, Chapman D, Amass L, Grogan M; THAOS Investigators. Temporal Trends of Wild-Type Transthyretin Amyloid Cardiomyopathy in the Transthyretin Amyloidosis Outcomes Survey. JACC CardioOncol. 2021 Oct 19;3(4):537-546. doi: 10.1016/j.jaccao.2021.08.009. eCollection 2021 Oct. PMID 34729526
- [Derived] Gonzalez-Moreno J, Losada-Lopez I, Cisneros-Barroso E, Garcia-Pavia P, Gonzalez-Costello J, Munoz-Beamud F, Campistol JM, Fernandez-Torron R, Chapman D, Amass L. A Descriptive Analysis of ATTR Amyloidosis in Spain from the Transthyretin Amyloidosis Outcomes Survey. Neurol Ther. 2021 Dec;10(2):833-845. doi: 10.1007/s40120-021-00267-y. Epub 2021 Jul 30. PMID 34331265
- [Derived] Gentile L, Tournev I, Amass L, Chapman D, Mazzeo A; THAOS investigators. Phenotypic Differences of Glu89Gln Genotype in ATTR Amyloidosis From Endemic Loci: Update From THAOS. Cardiol Ther. 2021 Dec;10(2):481-490. doi: 10.1007/s40119-021-00226-6. Epub 2021 Jun 19. PMID 34148211
- [Derived] Waddington-Cruz M, Wixner J, Amass L, Kiszko J, Chapman D, Ando Y; THAOS investigators. Characteristics of Patients with Late- vs. Early-Onset Val30Met Transthyretin Amyloidosis from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Neurol Ther. 2021 Dec;10(2):753-766. doi: 10.1007/s40120-021-00258-z. Epub 2021 May 22. PMID 34024024
- [Derived] Gonzalez-Duarte A, Barroso F, Mundayat R, Shapiro B. Blood pressure and orthostatic hypotension as measures of autonomic dysfunction in patients from the transthyretin amyloidosis outcomes survey (THAOS). Auton Neurosci. 2019 Dec;222:102590. doi: 10.1016/j.autneu.2019.102590. Epub 2019 Oct 23. PMID 31726319
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- [Derived] Pinto MV, Pinto LF, Dias M, Rosa RS, Mundayat R, Pedrosa RC, Waddington-Cruz M. Late-onset hereditary ATTR V30M amyloidosis with polyneuropathy: Characterization of Brazilian subjects from the THAOS registry. J Neurol Sci. 2019 Aug 15;403:1-6. doi: 10.1016/j.jns.2019.05.030. Epub 2019 May 28. PMID 31163298
- [Derived] Damy T, Kristen AV, Suhr OB, Maurer MS, Plante-Bordeneuve V, Yu CR, Ong ML, Coelho T, Rapezzi C; THAOS Investigators. Transthyretin cardiac amyloidosis in continental Western Europe: an insight through the Transthyretin Amyloidosis Outcomes Survey (THAOS). Eur Heart J. 2022 Feb 3;43(5):391-400. doi: 10.1093/eurheartj/ehz173. PMID 30938420
- [Derived] Cruz MW, Pinto MV, Pinto LF, Gervais R, Dias M, Perez C, Mundayat R, Ong ML, Pedrosa RC, Foguel D. Baseline disease characteristics in Brazilian patients enrolled in Transthyretin Amyloidosis Outcome Survey (THAOS). Arq Neuropsiquiatr. 2019 Feb;77(2):96-100. doi: 10.1590/0004-282X20180156. PMID 30810593
- [Derived] Rubin J, Steidley DE, Carlsson M, Ong ML, Maurer MS. Myocardial Contraction Fraction by M-Mode Echocardiography Is Superior to Ejection Fraction in Predicting Mortality in Transthyretin Amyloidosis. J Card Fail. 2018 Aug;24(8):504-511. doi: 10.1016/j.cardfail.2018.07.001. Epub 2018 Aug 17. PMID 30010028
- [Derived] Mundayat R, Stewart M, Alvir J, Short S, Ong ML, Keohane D, Rill D, Sultan MB. Positive Effectiveness of Tafamidis in Delaying Disease Progression in Transthyretin Familial Amyloid Polyneuropathy up to 2 Years: An Analysis from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Neurol Ther. 2018 Jun;7(1):87-101. doi: 10.1007/s40120-018-0097-9. Epub 2018 Apr 9. PMID 29633228
- [Derived] Kristen AV, Maurer MS, Rapezzi C, Mundayat R, Suhr OB, Damy T; THAOS investigators. Impact of genotype and phenotype on cardiac biomarkers in patients with transthyretin amyloidosis - Report from the Transthyretin Amyloidosis Outcome Survey (THAOS). PLoS One. 2017 Apr 6;12(4):e0173086. doi: 10.1371/journal.pone.0173086. eCollection 2017. PMID 28384285
- [Derived] Maurer MS, Hanna M, Grogan M, Dispenzieri A, Witteles R, Drachman B, Judge DP, Lenihan DJ, Gottlieb SS, Shah SJ, Steidley DE, Ventura H, Murali S, Silver MA, Jacoby D, Fedson S, Hummel SL, Kristen AV, Damy T, Plante-Bordeneuve V, Coelho T, Mundayat R, Suhr OB, Waddington Cruz M, Rapezzi C; THAOS Investigators. Genotype and Phenotype of Transthyretin Cardiac Amyloidosis: THAOS (Transthyretin Amyloid Outcome Survey). J Am Coll Cardiol. 2016 Jul 12;68(2):161-72. doi: 10.1016/j.jacc.2016.03.596. PMID 27386769
- [Derived] Damy T, Maurer MS, Rapezzi C, Plante-Bordeneuve V, Karayal ON, Mundayat R, Suhr OB, Kristen AV. Clinical, ECG and echocardiographic clues to the diagnosis of TTR-related cardiomyopathy. Open Heart. 2016 Feb 8;3(1):e000289. doi: 10.1136/openhrt-2015-000289. eCollection 2016. PMID 26870387
- [Derived] Coelho T, Maurer MS, Suhr OB. THAOS - The Transthyretin Amyloidosis Outcomes Survey: initial report on clinical manifestations in patients with hereditary and wild-type transthyretin amyloidosis. Curr Med Res Opin. 2013 Jan;29(1):63-76. doi: 10.1185/03007995.2012.754348. Epub 2012 Dec 13. PMID 23193944
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461001&StudyName=Transthyretin-Associated%20Amyloidoses%20Outcome%20Survey%20%28THAOS%29%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: THAOS (Transthyretin Amyloidosis Outcome Survey) was a non-interventional, longitudinal observational survey opened to all participants with ATTR (Transthyretin Amyloidosis), including both inherited and wild-type forms of disease and those with TTR gene mutations without disease diagnosis. There was no planned enroll number. THAOS did not involve the administration of an intervention. Participants continued to receive their previous medications and all other standard care for their disease.
Groups:
- Tafamidis 20 mg Treated: All available data from participants who received Tafamidis 20 mg throughout the study.
- Tafamidis 61/80 mg Treated-Overall: All available data from participants who received Tafamidis 61/80 mg (Tafamidis 61mg/tafamidis meglumine 80 mg) throughout the study.
- Tafamidis 20 mg to 61/80 mg Treated-Overall: All available data from participants who received Tafamidis 20 mg but switched to 61/80 mg during the study.
- Tafamidis Other Treated-Overall: All available data from participants who received any other dose of Tafamidis throughout the study.
- Tafamidis Untreated: All available data from participants who had been enrolled in THAOS, signed the informed consent and who had not received tafamidis during the THAOS study.
Period: Overall Study
Arm/Group | Tafamidis 20 mg Treated | Tafamidis 61/80 mg Treated-Overall | Tafamidis 20 mg to 61/80 mg Treated-Overall | Tafamidis Other Treated-Overall | Tafamidis Untreated
Started | 1648 | 662 | 196 | 15 | 4197
Completed | 4 | 0 | 1 | 0 | 8
Not Completed | 1644 | 662 | 195 | 15 | 4189
Not completed — Withdrawal by Subject | 63 | 3 | 9 | 2 | 69
Not completed — Does not meet inclusion criteria | 0 | 12 | 0 | 0 | 18
Not completed — Participation in an interventional clinical trial | 81 | 4 | 7 | 0 | 63
Not completed — Physician Decision | 8 | 4 | 3 | 0 | 30
Not completed — Lost to Follow-up | 109 | 7 | 7 | 0 | 498
Not completed — Death | 197 | 81 | 12 | 4 | 939
Not completed — Participant transferred to another THAOS site | 6 | 0 | 0 | 0 | 7
Not completed — Participant moved out of the area, but did not transfer to another THAOS site | 37 | 29 | 46 | 0 | 91
Not completed — Site closure | 152 | 146 | 6 | 8 | 691
Not completed — Duplicate participant | 0 | 0 | 0 | 0 | 1
Not completed — Missing | 4 | 3 | 0 | 0 | 10
Not completed — Othe reasons | 987 | 373 | 105 | 1 | 1772

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who had been enrolled in THAOS study, signed the informed consent form, and either received doses of Tafamidis (presented by dose group) during the study or never received Tafamidis throughout the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafamidis 20 mg Treated | Tafamidis 61/80 mg Treated-Overall | Tafamidis 20 mg to 61/80 mg Treated-Overall | Tafamidis Other Treated-Overall | Tafamidis Untreated | Total
Number analyzed (Participants) | 1648 | 662 | 196 | 15 | 4197 | 6718
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at enrollment
  Years | 50.8 (17.75) | 76.0 (8.65) | 77.7 (10.66) | 77.9 (11.33) | 57.1 (19.08) | 58.1 (19.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 734 | 62 | 33 | 4 | 1581 | 2414
  Male | 914 | 600 | 163 | 11 | 2616 | 4304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Afro-Caribbean | 0 | 2 | 0 | 0 | 22 | 24
  American Hispanic | 8 | 4 | 0 | 1 | 16 | 29
  Asian | 110 | 12 | 3 | 0 | 170 | 295
  Black or African American | 11 | 53 | 3 | 2 | 225 | 294
  Caucasian | 600 | 512 | 46 | 12 | 2271 | 3441
  Latino American | 42 | 2 | 0 | 0 | 138 | 182
  Other | 18 | 0 | 1 | 0 | 113 | 132
  Missing | 859 | 77 | 143 | 0 | 1242 | 2321

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who administered a medicinal product without regard to possibility of causal relationship with the study treatment. SAE was defined as one of the following: resulted in death; was life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); constituted a congenital anomaly/birth defect. Treatment-emergent AE was defined as an AE with onset date occurring during the on-treatment period. AEs included all SAEs and non-SAEs.
Time Frame: From the start of data collection at Baseline (Day 1) to the end of data collection (Up to 14.4 years)
Population: TEAEs and SAEs were summarised for only Tafamidis treated set: all available data from participants who have been enrolled in THAOS, signed the informed consent and were on tafamidis treatment on or prior to the date of enrollment of THAOS, or subsequently initiated tafamidis treatment after the enrollment of THAOS.
Measure: Count of Participants; unit: Participants
Groups:
- Tafamidis 20 mg Treated-Overall: All available data from participants who received Tafamidis 20 mg throughout the study.
Arm/Group | Tafamidis 20 mg Treated-Overall | Tafamidis 61/80 mg Treated-Overall | Tafamidis 20 mg to 61/80 mg Treated-Overall | Tafamidis Other Treated-Overall
Number analyzed (Participants) | 1648 | 662 | 196 | 15
Participants
  Participants with Adverse Events | 621 | 175 | 66 | 4
  Participants with Serious Adverse Events | 331 | 138 | 41 | 3

2. Primary Outcome: Number of Participants With Treatment Emergent Treatment Related AEs and SAEs
Description: A treatment-related AE was any untoward medical occurrence attributed to the administered medicinal product in a participant who received study drug. Treatment emergent AEs included both SAEs and all non-SAEs. A treatment-related SAE was a treatment-related AE and was defined as any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); constituted a congenital anomaly/birth defect. Causality was assessed by the investigator.
Time Frame: From the start of data collection at Baseline (Day 1) to the end of data collection (Up to 14.4 years)
Population: Treatment emergent treatment related AEs and SAEs were summarised for only tafamidis treated set: all available data from participants who have been enrolled in THAOS, signed the informed consent and were on tafamidis treatment on or prior to the date of enrollment of THAOS, or subsequently initiated tafamidis treatment after the enrollment of THAOS.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg Treated-Overall | Tafamidis 61/80 mg Treated-Overall | Tafamidis 20 mg to 61/80 mg Treated-Overall | Tafamidis Other Treated-Overall
Number analyzed (Participants) | 1648 | 662 | 196 | 15
Participants
  Participants with Adverse Events | 47 | 11 | 1 | 2
  Participants with Serious Adverse Events | 28 | 5 | 0 | 1

3. Primary Outcome: Number of All-Cause Deaths
Description: Number of deaths due to any cause was analyzed as time from enrollment or first treatment of tafamidis.
Time Frame: From the start of data collection at Baseline (Day 1) to the end of data collection (Up to 14.4 years)
Population: Tafamidis treated set included participants who were on tafamidis at or prior to the enrollment, as well as participants who were not on tafamidis at enrollment but subsequently initiated tafamidis treatment during the study. Tafamidis untreated set included participants who were enrolled and never received tafamidis throughout the study, as well as participants who were not on tafamidis before or at enrollment but subsequently initiated tafamidis treatment during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Tafamidis Treated-Overall: All available data from participants who had been enrolled in THAOS, signed the informed consent and who received tafamidis treatment on or prior to the date of enrollment in THAOS. All available data from first dose of tafamidis until final treatment discontinuation of tafamidis or end of follow-up in THAOS (whichever was earlier) for participant who received tafamidis at the time of enrollment in THAOS but subsequently initiated treatment with tafamidis. For outcome measures, a participant could be reported in both the tafamidis untreated and tafamidis treated sets if the participant initiated treatment with tafamidis after beginning participation in THAOS.
- Tafamidis Untreated-Overall: All available data from participants who had been enrolled in THAOS, signed the informed consent and who had not received tafamidis during the THAOS study; and for those participants who were not on tafamidis during or after initial enrollment in THAOS but then started receiving tafamidis post enrollment, all available data collected before receiving the first dose of tafamidis while in THAOS. Available data after a participant discontinued treatment with tafamidis were excluded.
Arm/Group | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 2521 | 5686
Participants | 158 | 1038

4. Secondary Outcome: Number of Participants With Modified Polyneuropathy Disability (mPND) Scores at Baseline
Description: Modified Polyneuropathy Disability (mPND) is a score that categorizes participants into six stages (0, I,II, IIIa, IIIb, IV) based on mobility status. 0 = No sensory disturbances in the feet and able to walk without difficulty; I=Sensory disturbances in the feet but able to walk without difficulty; II=Some difficulties with walking but can walk without aid; IIIa=Able to walk with 1 stick or crutch; IIIb=Able to walk with 2 sticks or crutches; IV=Not ambulatory, confined to a wheelchair or bedridden. Higher stage indicates lower mobility status.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: Overall analysis set:all enrolled participants in THAOS study.Tafamidis treated set:participants who were on tafamidis at or prior to the enrollment, as well as those who were not on tafamidis at enrollment but subsequently received tafamidis during the study.Tafamidis untreated set:participants who were enrolled and never received tafamidis throughout the study, as well as those who were not on tafamidis before or at enrollment but subsequently started tafamidis treatment during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All enrolled participants in THAOS study.
  Note：for outcome measures, a participant could be reported in both the tafamidis untreated and tafamidis treated sets if the participant initiated treatment with tafamidis after beginning participation in THAOS.
- Tafamidis Treated-Overall: All available data from participants who had been enrolled in THAOS, signed the informed consent and who received tafamidis treatment on or prior to the date of enrollment in THAOS. All available data from first dose of tafamidis until final treatment discontinuation of tafamidis or end of follow-up in THAOS (whichever was earlier) for participant who received tafamidis at the time of enrollment in THAOS but subsequently initiated treatment with tafamidis. For outcome measures, a participant could be considered part of both the tafamidis untreated and tafamidis treated sets if the participant initiated treatment with tafamidis after beginning participation in THAOS.
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4434 | 1689 | 3785
Participants
  0 | 1860 | 512 | 1731
  I | 1642 | 785 | 1372
  II | 492 | 255 | 349
  IIIa | 226 | 84 | 160
  IIIb | 136 | 37 | 106
  IV | 78 | 16 | 67

5. Secondary Outcome: Number of Participants With Coutinho Disease Stages at Baseline
Description: Coutinho disease stages is the most common classification used to capture ATTR (Transthyretin Amyloidosis) disease progression. Participants with stage 0 disease are asymptomatic, Participants with stage 1 (mild) disease are ambulatory, Participants with stage 2 (moderate) disease are ambulatory but require assistance and/or have involvement of the upper limbs, and Participants with stage 3 (severe) disease are bedridden or wheelchair-bound.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4434 | 1689 | 3785
Participants
  Stage 0 | 1860 | 512 | 1731
  Stage 1 | 2134 | 1040 | 1721
  Stage 2 | 362 | 121 | 266
  Stage 3 | 78 | 16 | 67

6. Secondary Outcome: Number of Participants With Karnofsky Performance Index at Baseline
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky performance score is 10 level score which ranges between 10 (moribund) to 100 (normal, no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All enrolled participants in THAOS study.
  Note：for outcome measures, a participant could reported in both the tafamidis untreated and tafamidis treated sets if the participant initiated treatment with tafamidis after beginning participation in THAOS.
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4764 | 1895 | 3998
Participants
  10 | 2 | 1 | 2
  20 | 6 | 0 | 6
  30 | 6 | 3 | 3
  40 | 82 | 15 | 71
  50 | 140 | 31 | 121
  60 | 271 | 92 | 209
  70 | 492 | 200 | 375
  80 | 944 | 436 | 728
  90 | 1127 | 633 | 890
  100 | 1694 | 484 | 1593

7. Secondary Outcome: Number of Participants With Heart Failure at Baseline
Description: Heart failure, also known as congestive heart failure is a cardiovascular event.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Participants | 2717 | 1125 | 2245

8. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Classifications at Baseline
Description: New York Health Association (NYHA) functional classification included: Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity; fatigue, palpitation, or dyspnea with ordinary physical activity), Class III (marked limitation of physical activity; fatigue, palpitation, or dyspnea with less than ordinary physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest).
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 2380 | 922 | 1963
Participants
  I | 304 | 133 | 252
  II | 1341 | 557 | 1088
  III | 664 | 222 | 556
  IV | 71 | 10 | 67

9. Secondary Outcome: Number of Participants Diagnosed With ATTR at Baseline
Description: Participants diagnosed with Transthyretin Amyloidosis (ATTR) at baseline with assessed category of yes, no, and unknown.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6035 | 2408 | 5046
Participants
  Yes | 4773 | 2368 | 3794
  No | 1234 | 36 | 1227
  Unknown | 28 | 4 | 25

10. Secondary Outcome: Number of Participants With Prior Misdiagnosis at Baseline
Description: Number of participants with ATTR and participants who had prior misdiagnosis at the baseline were reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Participants | 616 | 283 | 493

11. Secondary Outcome: Number of Participants With ATTR Genotypes at Baseline
Description: Genetic mutation leads to misfolding of protein transthyretin (TTR) which results in ATTR. In this outcome, number of participants with ATTRv mutation type and wild type TTR were reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Overall: All enrolled participants in THAOS study.
  Note: for outcome measures, a participant could be reported in both the tafamidis untreated and tafamidis treated sets if the participant initiated treatment with tafamidis after beginning participation in THAOS.
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Participants
  ATTRv mutation | 4950 | 1743 | 4365
  Wild type | 1768 | 778 | 1321

12. Secondary Outcome: Number of Participants With Past or Current Clinical Trial Participation at Baseline
Description: Number of participants had previous or current participant in any clinical trials at the baseline.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 5270 | 2149 | 4273
Participants
  Yes | 853 | 473 | 669
  No | 4417 | 1676 | 3604

13. Secondary Outcome: Number of Participants With Past or Current Tafamidis Compassionate Use/Early Access or Other Non-commercial Program at Baseline
Description: Number of participants being allowed for the use of Tafamidis when under strict conditions, Tafamidis was in development and made available to groups of participants who have a disease with no satisfactory authorised therapies and who cannot enter clinical trials.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 3267 | 1490 | 2461
Participants
  Yes | 85 | 80 | 38
  No | 3182 | 1410 | 2423

14. Secondary Outcome: Number of Participants With Known Family History of Symptomatic ATTR at Baseline
Description: Number of participants whether with family history of symptomatic ATTR amyloidosis at Baseline were reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6676 | 2513 | 5652
Participants
  Yes | 3874 | 1365 | 3485
  No | 2243 | 873 | 1792
  Unknown | 559 | 275 | 375

15. Secondary Outcome: Number of Affected Generations at Baseline
Description: The mean of affected generations in participants with a known family history was reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Generation
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 3730 | 1337 | 3344
Generation | 1.5 (0.95) | 1.5 (1.01) | 1.5 (0.96)

16. Secondary Outcome: Derived Neuropathy Impairment Score-Lower Limb (NIS-LL) at Baseline
Description: Neuropathy Impairment Score - Lower Limb (NIS-LL) assessed motor, sensory and reflex activity specifically in the lower limbs and combined total scores for the lower limbs were collected and reported. Derived NIS LL score extends from 0 (normal functions) to a maximum possible value of 88 points, the scale is additive for all deficits and is applied bilaterally for each modality tested: 1) muscle strength: 0 (normal)-4 (paralysis), higher score = more weakness; 2) sensory and 3) reflex testings: 0=normal, 1=decreased, or 2=absent. Reflex score: 0 (normal)-10 (present), higher score =present in more anatomic sites; Motor score: 0-160 (full range of motion with maximum resistance across all anatomical sites), higher score=more impairment. Sensory Score has a range of 0 to the normal value of 124 where ratings are coded as 0=absent; 1=decreased; 2=normal.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Score on a scale
  Derived NIS-LL Score: number analyzed (Participants) | 2969 | 1035 | 2686
  Derived NIS-LL Score | 14.0 (20.73) | 20.3 (20.17) | 12.7 (20.14)
  Reflex Score: number analyzed (Participants) | 3995 | 1355 | 3569
  Reflex Score | 8.2 (3.05) | 7.5 (3.13) | 8.3 (2.94)
  Motor Score: number analyzed (Participants) | 3857 | 1406 | 3427
  Motor Score | 152.2 (19.11) | 150.6 (18.98) | 152.8 (18.41)
  Sensory Score: number analyzed (Participants) | 2670 | 836 | 2473
  Sensory Score | 108.2 (25.83) | 97.6 (26.79) | 109.4 (25.19)

17. Secondary Outcome: Body Mass Index (BMI) at Baseline
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6512 | 2485 | 5494
kg/m^2 | 26.3 (17.93) | 26.5 (24.14) | 25.9 (11.12)

18. Secondary Outcome: Modified Body Mass Index (mBMI) at Baseline
Description: mBMI was calculated by multiplying BMI by serum albumin levels [gram/liter (g/L)]. mBMI was measured as kg/m^2*g/L. A progressive decline in mBMI indicated worsening of disease severity.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (kg/m^2)*(g/L)
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4370 | 1846 | 3672
(kg/m^2)*(g/L) | 1078 (240.9) | 1063.1 (228.8) | 1083.3 (242.4)

19. Secondary Outcome: Sitting Systolic and Diastolic Blood Pressures (SBP and DBP) at Baseline
Description: BP (Blood Pressure) is the pressure of the blood within the arteries. It is produced primarily by the contraction of the heart muscle. BP measurement is recorded by 2 numbers: systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles). Available sitting SBP and DBP at Baseline were reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: Overall:all available data from enrolled participants.Tafamidis treated:available data from enrolled participants that were on tafamidis at or prior to the enrollment,and those not on tafamidis at the enrollment but later initiated tafamidis.Tafamidis untreated:available data from enrolled participants and did not receive tafamidis throughout and those not on tafamidis prior or at enrollment but later initiated tafamidis.Number analyzed=participants with available BP data collected at baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2473 | 5686
mmHg
  Sitting Systolic BP (mmHg): number analyzed (Participants) | 6490 | 2473 | 5475
  Sitting Systolic BP (mmHg) | 123.7 (18.67) | 125.3 (18.78) | 122.9 (18.15)
  Sitting Diastolic BP (mmHg): number analyzed (Participants) | 6487 | 2473 | 5472
  Sitting Diastolic BP (mmHg) | 75.3 (11.69) | 75.6 (11.56) | 75.1 (11.58)

20. Secondary Outcome: Left Ventricular (LV) Septum Thickness at Baseline
Description: Cardiac amyloidosis is attributable to intramyocardial amyloid infiltration, which leads to a progressive increase of ventricular wall thickness and stiffness. A left ventricular (LV) wall thickness ≥12 mm plus at least one red flag should raise the suspicion of cardiac amyloidosis.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: Overall analysis set: All available data from enrolled participants in THAOS study. Tafamidis treated set: All available data from participants enrolled in THAOS that were on tafamidis at and prior to the enrollment; participant not on tafamidis at the enrollment subsequently initiated treatment. Tafamidis untreated set: All available data from participants enrolled in THAOS and did not receive tafamidis during the study, including those initiated receiving tafamidis post enrollment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 3036 | 1298 | 2429
mm | 15.2 (5.27) | 15.3 (4.31) | 15.2 (5.52)

21. Secondary Outcome: Left Ventricular (LV) Ejection Fraction at Baseline
Description: Left ventricular dysfunction, a condition in which the left ventricle of the heart exhibits a decreased functionality, was assessed based on systolic ejection fraction. Systolic ejection fraction was the fraction of the end-diastolic volume (EDV) that was ejected out of left ventricle with each contraction.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 2907 | 1263 | 2301
Percentage | 53.6 (13.46) | 54.3 (12.61) | 53.5 (13.77)

22. Secondary Outcome: Euro Quality of Life-5 Dimensions-3 Level (EQ-5D-3L): Visual Analog Scale (VAS) Overall Health Score at Baseline
Description: EQ-5D-3L VAS: participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. The VAS component rated the current health state on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicating a better health state.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4478 | 1709 | 3910
Score on a scale | 71.0 (20.80) | 70.2 (20.01) | 71.7 (20.98)

23. Secondary Outcome: EQ-5D-3L: VAS Derived Index at Baseline
Description: The EQ-5D-3L VAS derived index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value. This corresponds to the best possible health status, the scale of the Derived Index is 0 [death] to 1 [perfect health]. EQ-5D-3L VAS overall health score and derived score data were sourced from different part of the EQ-5D questionnaire and are conceptually different from each other as EQ VAS is a 0-100 scale and EQ-5D index is a value attached to an EQ-5D profile according to a set of weights that reflect, on average, participant's preferences about how good or bad the state is. More data were collected for EQ-5D index score compared to EQ VAS overall health score at the baseline.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4550 | 1736 | 3969
Score on a scale | 0.8 (0.20) | 0.8 (0.19) | 0.8 (0.20)

24. Secondary Outcome: Norfolk Total Quality of Life (QoL) Score at Baseline
Description: Norfolk QOL: 35-item participant-rated questionnaire used to assess impact of neuropathy on the quality of life of participants diagnosed with ATTR. Scoring was based on 35 questions that yield a TQOL as well as 5 subscale scores: activities of daily living, large fiber neuropathy/physical functioning, small fiber neuropathy, autonomic neuropathy, and symptoms. TQOL= sum of all the items, total possible score range= -2 to 138, where higher score=worse quality of life.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 4605 | 1795 | 4002
Score on a scale | 24.3 (28.10) | 25.2 (27.30) | 23.1 (27.90)

25. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) at Baseline
Description: Following parameters were analyzed: heart rate, PR interval, QT interval, QRS interval and QT interval corrected using Fridericia's formula (QTcF). Abnormal findings in ECG were based on investigator's discretion.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Participants | 2911 | 1226 | 2315

26. Secondary Outcome: Number of Participants With Atrial Fibrillation/Flutter, Pacemaker Implanted, and Implantable Cardioverter/Defibrillator (ICD) at Baseline
Description: Number of participants with atrial fibrillation/flutter (rapid, irregular heart rhythm), implanted artificial cardiac pacemaker, and implantable cardioverter-defibrillator (ICD) (detects and stops irregular heartbeats, also called arrhythmias) were reported.
Time Frame: At the start of data collection at Baseline (Day 1)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Tafamidis Treated-Overall | Tafamidis Untreated-Overall
Number analyzed (Participants) | 6718 | 2521 | 5686
Participants
  Atrial Fibrillation/Flutter | 667 | 290 | 501
  Pacemaker Implanted | 364 | 167 | 266
  ICD Implanted | 127 | 62 | 99

ADVERSE EVENTS:
Time Frame: From the start of data collection at Baseline (Day 1) to the end of data collection (Up to 14.4 years)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Tafamidis 20 mg Treated-Overall | Tafamidis 61/80 mg Treated-Overall | Tafamidis 20 mg to 61/80 mg Treated-Overall | Tafamidis Other Treated-Overall | Tafamidis Untreated
All-Cause Mortality (participants affected / at risk) | 197/1648 | 81/662 | 12/196 | 4/15 | 939/4197
Serious Adverse Events (participants affected / at risk) | 333/1648 | 138/662 | 41/196 | 3/15 | 4/4197
Other Adverse Events (participants affected / at risk) | 94/1648 | 3/662 | 0/196 | 1/15 | 0/4197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tafamidis 20 mg Treated-Overall (N=1648) | Tafamidis 61/80 mg Treated-Overall (N=662) | Tafamidis 20 mg to 61/80 mg Treated-Overall (N=196) | Tafamidis Other Treated-Overall (N=15) | Tafamidis Untreated (N=4197)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Familial amyloidosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 3 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Amyloidosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 12 | 3 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pregnancy of partner (Social circumstances) | 8 | 0 | 0 | 0 | 0
Abdominal cavity drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0/15
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0/15
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0/15
Acute left ventricular failure (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 5 | 5 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 7 | 3 | 0 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 2 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 3 | 6 | 2 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Atrioventricular dissociation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac amyloidosis (Cardiac disorders) | 3 | 2 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 6 | 8 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 34 | 32 | 18 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 4 | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 15 | 14 | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiomyopathy acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Defect conduction intraventricular (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 2 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Sinoatrial block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Hypertrophic cardiomyopathyv (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 2 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 3 | 0 | 0 | 0
Death (General disorders) | 8 | 11 | 4 | 1 | 1
Disease progression (General disorders) | 8 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 16 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 3 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1 | 0 | 0
Multi-organ disorder (General disorders) | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 6 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 2 | 0 | 0 | 0 | 0
Biliary fistula (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 0 | 0 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 8 | 2 | 1 | 0 | 0
Chikungunya virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 5 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infective keratitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 8 | 0 | 0 | 0 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 13 | 6 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 8 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 10 | 2 | 2 | 0 | 0
Septic shock (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary bladder abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 12 | 1 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 5 | 2 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Complications of transplanted liver (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Liver transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Transplantation complication (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 3 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Enzyme abnormality (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 4 | 0 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 7 | 0 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 8 | 5 | 2 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 14 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 4 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 1 | 2 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Liver transplant (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 2 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Amyloidosis senile (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Heart transplant rejection (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg Treated-Overall (N=1648) | Tafamidis 61/80 mg Treated-Overall (N=662) | Tafamidis 20 mg to 61/80 mg Treated-Overall (N=196) | Tafamidis Other Treated-Overall (N=15) | Tafamidis Untreated (N=4197)
Urinary tract infection (Infections and infestations) | 94 | 3 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
A total of 6718 evaluable participants were enrolled in this study. The database has 6752 participants and the discrepancy in the numbers is due to 1 system screen failure and 33 subjects that are either duplicates or were transferred to a different site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT00628745/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT00628745/SAP_001.pdf